CLINICAL TRIAL: NCT06389591
Title: A Phase I Study of RNA-Lipid Particle (RNA-LP) Vaccines for Recurrent Adult Glioblastoma (GBM)
Brief Title: RNA-Lipid Particle (RNA-LP) Vaccines for Recurrent Adult Glioblastoma (GBM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202301957; R37CA251978 (NIH); OCR44973 (Other: University of Florida)
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Glioblastoma
Keywords: brain tumor; malignant brain tumor; immunotherapy; adult
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: pp65 RNA-LPs (DP1) before biopsy (Experimental): Participants will receive pp65 RNA-LPs (DP1) starting before tumor biopsy/resection. All patients will receive three pp65 RNA-LP vaccines (DP1) before receiving full dose monthly RNA-LPs (RNA loaded lipid particles, RNA-LPs, DP2).
  Interventions: Biological: pp65 RNA loaded lipid particles, pp65 RNA-LPs (Drug Product 1 or DP1); Biological: RNA loaded lipid particles, RNA-LPs (Drug Product 2 or DP2)

INTERVENTIONS:
Biological: pp65 RNA loaded lipid particles, pp65 RNA-LPs (Drug Product 1 or DP1) — pp65 RNA loaded lipid particles or pp65 RNA-LPs administered intravenously
Biological: RNA loaded lipid particles, RNA-LPs (Drug Product 2 or DP2) — personalized tumor mRNA, pp65 fl LAMP mRNA and DOTAP liposomes or RNA loaded lipid particles, RNA-LPs administered intravenously

SUMMARY:
This is a Phase I study to demonstrate the manufacturing feasibility and safety, and to determine the maximum tolerated dose (MTD) of RNA-LP vaccines in adult patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
This is a first in human Phase I study of RNA-LP vaccines for recurrent adult glioblastoma. Participants will receive two study drug products. The first, pp65 RNA-LP, is a messenger RNA (mRNA) pp65 vaccine given for the first 3 vaccines to try to change how the tumor behaves. The second study drug RNA-LP, given as monthly vaccines 4-15, includes pp65 mRNA and tumor RNA from each patient's tumor tissue.

Patients will may receive up to three pp65 RNA-LP vaccines (DP1) before receiving full dose monthly RNA-LPs (RNA loaded lipid particles, RNA-LPs, DP2). All participants will receive the same number of vaccines, up to 15.

The immunotherapy with RNA lipid particle (RNA-LP) vaccines is the treatment portion of this study. During this study, we will make, test and give the RNA-LP vaccine therapy. As part of this study, participants will undergo up to 4 additional MRIs.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18years
* Histopathologically proven GBM using the 2021 WHO Classification of Tumors of the CNS (WHO CNS5).
* Unequivocal evidence of tumor progression as documented by brain MRI scan per RANO criteria.
* Tumor must have a primary supratentorial component at the time of disease progression.
* Patients must have received surgery and and should have completed Fractionated Radiation therapy with concurrent temozolomide as frontline treatments for primary disease and be at least 12 weeks post chemoradiation completion.
* Patient must be at least 90 days from completion of prior radiation
* Any adverse events patient has experienced from prior therapy must have resolved to ≤ Gr. 1 according to CTCAE (NCI Common Terminology Criteria for Adverse Events) v5.0 prior to enrollment
* Patient must be either weaned off steroids or weaned onto physiologic dosing at the time of enrollment.
* Patient must be a candidate for surgery/biopsy as acceptable standard of care for sterile collection of tumor material in a manner suitable for RNA extraction, amplification, and loading of lipid particles (LPs).
* A diagnostic contrast-enhanced MRI of the brain must be performed preoperatively and postoperatively. Pre-op MRI must be performed within 28 days prior to study enrollment.
* Performance Score: (KPS) ≥ 60. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Bone Marrow:

  * ANC (Absolute neutrophil count) ≥ 1,500µl (unsupported)
  * Platelets ≥ 100/µl (unsupported for at least 3 days)
  * Hemoglobin > 8 g/dL
* Renal:

  * BUN ≤ 25 mg/dl
  * Creatinine ≤ 1.7 mg/dl
* Hepatic

  * Bilirubin ≤ 2.0 mg/dl
  * ALT ≤ 5 times institutional upper limits of normal for age
  * AST ≤ 5 times institutional upper limits of normal for age
* Patient must be able to give consent.
* For women of childbearing potential (WOCBP), negative serum/urine pregnancy test at enrollment.
* WOCBP must be willing to use acceptable contraceptive methods to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug.
* Males with female partners of childbearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.

Exclusion Criteria:

* Patients who received prior treatment with bevacizumab.
* Known active infection (requiring treatment by antiviral or antibiotics) or immunosuppressive disease.
* Patients with multifocal recurrent disease characterized by more than one enhancing lesion separated by noncontiguous T2/FLAIR signal abnormality. Patients with recurrence outside of the original tumor site are eligible if there is stability at the original site of disease.
* Patients with uncontrolled seizure disorders
* Any patients that have received any live vaccines within 30 days prior to enrollment
* Tumors with primary localization to the brainstem or spinal cord
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization.
  * Unstable cardiac arrhythmias, abnormalities, or transmural myocardial infarction within the last 6 months.
  * Acute bacterial or fungal infection requiring intravenous treatment at study treatment.
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at study treatment
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
  * Patients with autoimmune disease requiring medical management with immunosuppressants.
  * Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy.
  * Pregnancy or women of childbearing potential and men who are sexually active and who are unwilling or unable to use an acceptable method of contraception for the entire study period; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Women of childbearing potential must not be pregnant or breast-feeding.
* Participants who are receiving any other investigational agents or who have been treated on any other therapeutic clinical protocols within 30 days prior to projected first dose of study treatment.
* Participants who are unwilling or unable to receive treatment and undergo follow-up evaluations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of vaccines meeting release criteria in the DLT window during the first three vaccines | from the date of surgery until administration of third vaccine, up to 20 weeks
  Manufacturing feasibility will be determined based on the percentage of vaccines that are successfully manufactured in the DLT window during the first three vaccines. If two-thirds of vaccines are successfully manufactured with Qa/Qc clearance, the investigators will conclude that RNA-LPs can be successfully manufactured.
Incidence of investigational treatment related toxicities | from first vaccine to 30 days after last dose of vaccine administered, up to 17 months
  AEs and SAEs must be reported begins at time of first investigational product is received and ends 30 days after last investigational product is given.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ghiaseddin, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

REFERENCES:
- [Derived] Carrera-Justiz S, Aghaee M, Qdaisat S, Weidert F, Garcia GA, Fagman L, Zhang D, Stover B, Moor RSF, Xie C, Goldenberg E, von Roemeling C, Doonan B, Chardon-Robles J, Elliott L, Sawyer WG, Deleyrolle LP, Sahay B, Foster TP, Seligson ND, Rahman M, Ghiaseddin A, Castillo P, Lee JH, Silver NL, Doty A, Ligon JA, Milner RJ, Mitchell D, Mendez-Gomez H, Moore H, Sayour EJ. Systemic mRNA vaccines elicit rapid immune activation in canine brain tumors. J Immunother Cancer. 2025 Nov 11;13(11):e011817. doi: 10.1136/jitc-2025-011817. PMID 41218853
- [Derived] Villanueva MT. RNA delivery heats up cold tumours. Nat Rev Drug Discov. 2024 Jul;23(7):497. doi: 10.1038/d41573-024-00098-0. No abstract available. PMID 38858569